CLINICAL TRIAL: NCT03905889
Title: Targeting PIM1 and CDK4/6 Kinases in Renal Cell Carcinoma (PICKRCC): A Phase Ib Study of Abemaciclib (VerzenioTM) in Combination With Sunitinib in Metastatic Renal Cell Carcinoma
Brief Title: A Study of Abemaciclib in Combination With Sunitinib in Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Brown University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 411
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Carcinoma Metastatic
Keywords: Renal cell carcinoma; Abemaciclib; Sunitinib
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — abemaciclib; Sunitinib

STUDY DESIGN:
Intervention Model Description: This is a single-arm, non-randomized prospective phase Ib study with expansion. The goal is to determine the maximal tolerated dose by assessing dose limiting toxicities. A classic "3+3" design is used. There are a total of 3 dose levels (level -1, 1, and 2) with dose level 1 as the starting dose. Once the maximum tolerated dose is established, a cohort of an additional 10 subjects will be enrolled at the established dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experimental Abemaciclib and Sunitinib (Experimental): For the dose escalation phase, Subjects will receive a 21-day cycle of continuous oral daily Sunitinib in combination with Abemaciclib every 12 hours for 14 days followed by 7 days off. Using a traditional 3 x 3 study design assessing dose limiting toxicity, if the initial prescribed dosing of these 2 medications (Dose Level 1) is tolerated by the first 3 subjects, the study will pause for a 30 day time period between cohorts to assess toxicity. If no dose limiting toxicity is identified, the next cohort of 3 new subjects will be treated at the next higher dose level (Dose Level 2). If the original cohort treated at Dose Level 1 do not tolerate the combination of medications, the medication regimen will be modified to a lower dose (Dose Level - 1). A dose expansion phase is included which will evaluate the combination of Abemaciclib in combination with Sunitinib when given at the maximum tolerated dose as determined from the from dose escalation phase.
  Interventions: Drug: Abemaciclib; Drug: Sunitinib

INTERVENTIONS:
Drug: Abemaciclib — Subjects will by given oral Abemaciclib every 12 hours for 14 days followed by 7 days off (i.e. a 21 day cycle). The initial dose will be 100 mg (Dose level 1) followed by 150 mg (Dose Level 2) depending on tolerability and toxicity assessment of the combination of medications. If at Dose Level 1 subjects cannot tolerate the combination of medications, the Abemaciclib would not be increased, and the dose will remain stable at 100 mg (Dose Level -1).
  Other Names: Verzenio
Drug: Sunitinib — Subjects will take oral Sunitinib daily for the 21-day cycle. Dosing will be at 50 mg for both Dose Levels 1 and 2. If the combination of the 2 medications is not tolerated by Subjects at Dose Levels 1 a lower dose of Sunitinib (37.5 mg) will be given (Dose Level -1).
  Other Names: Sutent

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and maximal tolerated dose (MTD) of the combination of Abemaciclib and Sunitinib administered orally in patients with advanced and metastatic renal cell carcinoma. This study consists of two parts: Dose Escalation and Dose Expansion. During the dose escalation phase, participants will be sequentially enrolled in a standard 3 x 3 dose escalation study design to receive oral Abemaciclib in Combination with Sunitinib. The purpose of this dose escalation is to determine the maximal tolerated dose based on assessment of any dose limiting toxicity. The Dose Expansion Phase will enroll additional participants at the established maximal tolerated dose to further evaluate safety, tolerability, as well as the pharmacokinetics and pharmacodynamics of this combination drug regimen.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) accounted for about 64, 000 new cancer diagnoses in the USA in 2018. Up to 30% of those diagnoses will be patients with metastatic disease. Additionally, up to 50% of patients who undergo partial or radical nephrectomy will develop metastatic disease.. There is no cure for metastatic RCC, thus, metastatic RCC represents a significant cancer burden. Numerous directed therapies are available to improve overall survival but these do not result in durable complete responses. However, recent pre-clinical studies of RCC have demonstrated that Abemaciclib, a CDK4/6 and PIM1 kinase inhibitor, induces rapid, dramatic, and sustained tumor regression when used in combination with Sunitinib.

Our objectives for this study are as follows:

Primary Objectives:

* Determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of the combination of Abemaciclib with Sunitinib for patients with metastatic renal cell carcinoma. Additionally, determine pharmacokinetics (serum trough levels) of Abemaciclib and Sunitinib at steady state.
* Continued safety assessment of the combination of Abemaciclib and Sunitinib at the established maximum tolerated dose (i.e. the recommended Phase II dose)

Secondary Objectives:

Determine any anti-tumor activity in the dose expansion phase of the study. Tumor related activity will be assessed by:

* Length of progression free survival
* Disease response rate
* Time to disease response
* Disease control rate
* Duration of response
* Overall survival and progression free survival

ELIGIBILITY:
Inclusion Criteria:

1. Has histologic or cytologic evidence of metastatic renal cell carcinoma with histology predominantly (>50%) clear cell renal cell carcinoma solid neoplasm.
2. Has evidence of metastatic disease. Intermediate and poor risk patients according to International Metastatic Renal Cell Carcinoma Database criteria (IMDC) must have received prior combination ipilimumab and nivolumab therapy and subsequently experienced disease progression, or been offered ipilimumab and nivolumab combination therapy and refused, or be ineligible for combination ipilimumab and nivolumab therapy. Patients with favorable risk disease have no eligibility requirement for prior use of ipilimumab and nivolumab immunotherapy.
3. Intermediate and poor risk patients (according to IMDC criteria) must also have received prior cabozantinib therapy and subsequently experienced disease progression, or been offered cabozantinib therapy and refused, or be ineligible for cabozantinib therapy. Patients with favorable risk disease have no eligibility requirement for prior use of cabozantinib. Cytoreductive nephrectomy is allowed but not mandatory.
4. Has in the opinion of the investigator, a predicted life expectancy of more than 3 months.
5. Has presence of at least 1 lesion that is measurable or evaluable using RECIST v1.1. This is defined in at least one dimension as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT, MRI or calipers by clinical exam
6. Has either archival tissue for analysis or will require confirmation of disease with fresh biopsy. Tissue will not be required pre/post treatment for biomarker analysis.
7. Has an Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2.
8. Patients with central nervous system metastases must have received surgical and/or radiation treatment, the metastases must be neurologically stable, and patients must be off corticosteroids or receiving a stable low-dose regimen of corticosteroids (i.e., a daily dose of 10 mg or less of prednisone or equivalent) for at least 4 weeks prior to the first dose of study drug.
9. Has completed any prior anticancer treatment and must have recovered from any acute toxicities. The period between the last dose of prior treatment and the first dose of study drug treatment must be at least 1 week for radiotherapy, at least 3-4 weeks from prior VEGFR/mTOR/ or immunotherapy or any other tyrosine kinase inhibitor (TKI) therapy, and at least 4 weeks for treatment with investigational drugs
10. Must be able to swallow capsules and tablets.
11. Has adequate organ function (i.e. lung, liver, kidney, bone marrow), as evidenced by multiple laboratory value results within specific parameters.
12. Women of childbearing potential (WOCP) as defined as not surgically sterile or not postmenopausal) must have a negative result for a serum pregnancy test before study drug administration on cycle 1 day 1. WOCP must use a medically accepted method of contraception and must agree to continue use this method for the duration of the study and for 30 days after discontinuation of study drug.
13. If male, is surgically sterile, or, if capable of producing offspring, is currently using an approved method of birth control and agrees to continued use of this method for the duration of the study (and for 30 days after taking the last dose of study drug because of the possible effects on spermatogenesis).

Exclusion Criteria:

1. Predominately non-clear cell renal cell carcinoma histology (i.e. >50%)
2. Has had chemotherapy within 4 weeks or radiotherapy within 1 week prior to first dose of study drug or those who have not recovered from toxicities due to agents administered more than 4 weeks earlier.
3. Has ongoing or active infection requiring parenteral antibiotics.
4. Has uncontrolled hypertension despite adequate therapy (i.e., systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 90 mm Hg found on 2 separate occasions separated by 1 week).
5. Has diabetes mellitus with occurrence of more than 2 episodes of ketoacidosis in the 12 months prior to the first dose of study drug.
6. Has an active second malignancy other than curatively resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or other cancers for which they are treated with curative intent, and no known active disease in the 3 years prior to enrollment.
7. Has a primary brain tumor or has brain metastases from a non-renal cell cancer.
8. Has a QTcF interval greater than 470 msec, has a known history of QTcF prolongation, or has a history of torsade de pointes.
9. Has a known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C.
10. Has a known history of pulmonary fibrosis or any other restrictive lung disorder.
11. Has any other concurrent conditions including a medical, psychiatric, or social condition that, in the opinion of the investigator, could preclude the patient's participation in the study, pose an undue medical hazard, or interfere with the interpretation of the study results, including, but not limited to, patients with congestive heart failure (New York Heart Association [NYHA] Class III or IV), cardiac arrhythmia, or acute coronary syndromes within 6 months of enrollment.
12. Has used an investigational drug within 4 weeks prior to first dose of study drug or is currently participating in another investigational study.
13. Has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery or bariatric surgery).
14. Has a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Abemaciclib or Sunitinib.
15. Has previous use of a CDK4/6 kinase inhibitor (eg. ribociclib, palbociclib)
16. Has previous use of a PIM1 kinase inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | At the end of Cycle 1 (each cycle is 21 days)
  A standard 3+3 trial design will be used to determine the safest maximal tolerated dose of the combination of Abemaciclib with Sunitinib. Doses of each medication will be increased or decreased based on upon tolerability and assessment of any dose limiting toxicity(ies) that may occur in study subjects. Safety and toxicity will be evaluated using the NCI Common Toxicity Criteria.
Continued Toxicity assessment of the maximum tolerated dose (i.e the recommended Phase II dose) of Abemaciclib and Sunitinib as determined from the from dose escalation phase. | 44 days after the last dose of study drug
  Continued safety assessment of the combination of Abemaciclib and Sunitinib when administered at the maximal tolerated dose (i.e. the recommended phase 2 dose)
Pharmacokinetic Assessment of Abemaciclib and Sunitinib trough levels at steady state | Days 8, 15, 21, 28, 35, 42, 56, 63, 77, 84, 98 (at the beginning and weekly during cycles 1 and 2, days 1 and 15 of cycles 3-5; a cycle is 21-days)
  Assessment of steady state trough levels of Abemaciclib and Sunitinib

SECONDARY OUTCOMES:
Disease Control Rate | 54 weeks
  The number of subjects achieving a response (complete response, partial response, stable disease) on the combination regimen of Abemaciclib and Sunitinib at 6, 12, 24, 36, 45, and 54 weeks post initiation of treatment.
Progression Free Survival | 3 years
  The duration of time from the date of start of treatment until the criteria for disease progression is met by RECIST v1.1 criteria.
Overall Survival | 3 years
  Overall Survival rate from initiation of Abemaciclib and Sunitinib to completion of the protocol prescribed drug regimen and required follow up time period.
Median Progression Free Survival | 3 years
  The median number of days of progression free survival from initiation of Abemaciclib and Sunitinib to completion of the protocol prescribed drug regimen and required follow up time period.
Median Overall Survival | 3 years
  The median number of days of survival from initiation of Abemaciclib and Sunitinib to completion of the protocol prescribed drug regimen and required follow up time period.
Duration of Response | 3 years
  The period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Holder, MD, PhD, Principal Investigator — Lifespan Cancer Institute
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States